CLINICAL TRIAL: NCT01568645
Title: A Pilot Study of Treatment of Adults With Sickle Cell Disease Associated Pulmonary Hypertension Based on Hemodynamic Stratification: Safety and Tolerability Study of Imatinib and Carvedilol
Brief Title: Imatinib and Carvedilol for High Blood Pressure in the Lungs in Adults With Sickle Cell Disease
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 120093; 12-H-0093
Record Dates: First submitted 2012-03-30; First posted 2012-04-02 (Estimated); Last update posted 2018-07-05 (Actual); Status verified 2012-12-11

CONDITIONS: Pulmonary Hypertension
Keywords: Sickle Cell Anemia; Tyrosine Kinase Inhibitor; Platelet Derived Growth Factor; Beta Adrenergic Receptor Blocker; Pulmonary Vascular Disease; Sickle Cell Disease; Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary; Anemia, Sickle Cell | interventions — Carvedilol; Imatinib Mesylate

INTERVENTIONS:
Drug: Carvedilol
Drug: Imatinib

SUMMARY:
Background:

- About one-tenth of adults with sickle cell disease have pulmonary hypertension (high blood pressure in the lungs). This condition can cause shortness of breath, pain crisis, and congestive heart failure. It may even lead to death. Researchers want to test the drugs imatinib and carvedilol to see if they can treat high blood pressure in the lungs. Both drugs have been used to treat other types of heart problems, but they have not been tested as a treatment for high blood pressure related to sickle cell disease.

Objectives:

- To see if imatinib and carvedilol are safe and effective treatments for high blood pressure in the lungs in adults with sickle cell disease.

Eligibility:

- Adults at least 18 years of age who have sickle cell disease and have or may have high blood pressure in the lungs.

Design:

* Participants will be screened with a physical exam and medical history. They will also have different tests of heart and lung function, including a walking test and imaging studies. Blood and urine samples will also be collected.
* Participants who meet specific criteria will take one of two possible study drugs. Those who receive imatinib will take it daily. Those who receive carvedilol will take it twice a day.
* Participants will have weekly study visits for blood tests and other exams. The study drug dose will be adjusted at each weekly visit. It will be increased slowly to reach a target dose(based on the participant s weight) or to find a stable effective dose.
* Participants may continue to take their study drug for up to 24 weeks, with weekly study visits. Regular blood samples and heart and lung function tests will be performed.
* After 24 weeks, qualified participants may continue to take their study drug for up to 6 more months. They will have regular study visits to monitor the treatment.

DETAILED DESCRIPTION:
Sickle Cell Disease related pulmonary hypertension is a heterogeneous condition that results in a high mortality and for which no therapy has been documented to be beneficial. We propose to perform a safety and tolerability study of treatments based on right heart catheterization derived hemodynamic profiles associated with higher mortality in our cohort. These same hemodynamic profiles have previously been described and confirmed in other large cohorts as well. We propose treatment of sickle cell subjects with pulmonary arterial hypertension (PAH), defined hemodynamically by pulmonary arterial mean pressures (mPAP) of 25 mmHg or greater, with low estimated left ventricular filling pressures (low pulmonary capillary wedge pressures, or PCWP), and high pulmonary vascular resistance (PVR), with imatinib, a tyrosine kinase inhibitor that modifies the Platelet Derived Growth Factor (PDGF) pathway. PDGF is involved in Sickle Cell related PAH and there is now evidence that imatinib is effective in the treatment of idiopathic PAH. The hemodynamic profile of elevated mPAP with elevated left ventricular filling pressures is also associated with higher mortality rates, and we propose to treat this subgroup with carvedilol, a unique beta-adrenergic receptor antagonist that has been demonstrated to attenuate the adrenergic response and improve right and left heart function. The third subgroup with elevated mPAP is the hyperdynamic group, which by definition has low PVR and the absence of elevated left ventricular filling pressures. This group is also at higher risk but over a longer period of time and for less evident reasons. We will continue with aggressive sickle cell management in the hyperdynamic group according to the expertise offered by the Sickle Cell Group at the Clinical Center while systematically following them and intervening with optimal care. Those who do not quality for any of the three subgroups described above will go into a fourth subgroup and be followed for mortality and data sharing. Our primary endpoint is the safety and tolerability of these interventions and our secondary endpoints will be the clinical efficacy of these treatments.

ELIGIBILITY:
* Eligibility Criteria
* Subjects 18 years of age or older
* Must be able to provide written informed consent
* Subjects with SCD and prior RHC documenting mPAP greater than or equal to 25 mmHg
* Suspicion of Pulmonary Hypertension based on any of the below criterion:

<TAB>- exertional breathlessness

<TAB>- echocardiographic evidence of tricuspid insufficiency (TRVgreater than or equal to 2.7 m/s)

<TAB>- oxy-hemoglobin desaturation during six minute walking test

<TAB>- hypoxia requiring supplemental oxygen

<TAB>- pedal edema

<TAB>- ascites

<TAB>- elevated BNP

<TAB>- or history of acute chest syndrome, stroke, or other serious complication of vaso-occlusive disease

<TAB>- history of chest pain, syncopal events or thromboembolic events

<TAB>- The referring physician may refer the subject for other suspicious symptoms or findings of SCD-PH

INCLUSION CRITERIA:

Arm A (Imatinib)

1. Satisfaction of screening criteria
2. Subjects 18 years of age or older
3. Women of childbearing potential and male subjects must agree to use reliable methods of birth control (oral contraceptives, other hormonal contraceptives including vaginal contraceptive rings and contraceptive patches, barrier contraceptives such as condoms, an intra uterine device (IUD) or abstinence). This is because the effects of imatinib mesylate on the developing human fetus are not fully known.
4. Diagnosis of sickle cell disease (electrophoresis or HPLC)
5. Documentation of SS, SC, S-Beta thalassemia or other major sickling phenotypes)
6. Diagnosis of sickle cell disease associated pulmonary hypertension by right heart catheterization (mean PAP greater than or equal to 25 mmHg AND PCWP less than or equal to 15 mmHg with PVR greater than or equal to 3.0 Wood s Units)
7. WHO functional class II or III symptoms

Arm B (Carvedilol)

1. Satisfaction of screening criteria
2. Right heart catheterization (mean PAP greater than or equal to 25 mmHg AND PCWP > 15 mmHg
3. Clinically stable for at least 6 weeks prior to enrollment. PAH treatments must be stable for three months prior to study drug initiation. Prostacyclin analogs, type 5 phosphodiesterase inhibitors and endothelin-1 receptor antagonists are all allowed, alone or in combinations
4. Diagnosis of sickle cell disease (electrophoresis or HPLC documentation of SS, SC, S-Beta thalassemia or other major sickling phenotypes)
5. Women of childbearing potential and male subjects must agree to use reliable methods of birth control (oral contraceptives, other hormonal contraceptives including vaginal contraceptive rings and contraceptive patches, barrier contraceptives such as condoms, an intra uterine device (IUD) or abstinence). This is because the effects of Carvedilol in pregnancy is unknown (pregnancy risk factor C).
6. Subjects 18 years of age or older
7. WHO functional class II or III symptoms

Arm C (Hyperdynamic)

1. Sickle cell disease
2. Diagnosis of sickle cell disease associated pulmonary hypertension by right heart catheterization (mean PAP greater than or equal to 25 mmHg AND PCWP less than or equal to 15 mmHg with PVR < 3.0 Wood s Units)
3. Subjects 18 years of age or older

Arm D

1) Don t qualify for Arm A, B, or C after completing the baseline assessments.

EXCLUSION CRITERIA

Arm A (Imatinib):

1. Current pregnancy and lactation.
2. Life expectancy less than 6 months.
3. WHO functional class IV symptoms or NYHA-IV dyspnea.
4. Presence of any of the medical conditions that are considered to be the cause of subject s pulmonary hypertension by subject s physician, including but not limited to:

   <TAB>- Scleroderma.

   <TAB>- Known significant obstructive or restrictive respiratory disease with FEV1, FVC or TLC below 60 percent of predicted normal.

   <TAB>- Known diagnosis of Obesity-Hypoventilation Syndrome.

   <TAB>- Portal hypertension or Child Class B or C cirrhosis.

   <TAB>- Significant left ventricular dysfunction (LVEF below 50 percent), significant ischemic, valvular, constrictive or restrictive heart disease.
5. Persistently uncontrolled severe systemic hypertension (SBP above 160 mmHg or DBP above 100 mmHg)
6. Clinical diagnosis of decompensated congestive heart failure
7. Any initiation of new therapeutic intervention within the last 90 days or a dose change within 30 days, that is expected to have an impact on pulmonary hypertension, including but not limited to:

   1. <TAB>Specific pulmonary hypertension medication (e.g. prostacyclin analogues, endothelin receptor antagonists or phosphodiestrase-5 inhibitors)
   2. <TAB>Hydroxyurea
   3. <TAB>Scheduled blood transfusions or exchange transfusions
8. Any acute or chronic, physical or psychiatric impairment, likely to limit subject s ability to comply with study requirements as determined by investigators.
9. Subjects having inadequate organ function or hematopoeisis as defined below:

   1. Absolute Neutrophil Count (ANC) < 1200/mcL
   2. Platelets Count < 50, 000 / mcL
   3. ALT (SGPT) > 3 times upper limit of normal
   4. Creatinine greater than or equal to 2.0 mg/dl
   5. Creatinine Clearance < 60 mL/min/1.73 m sq
10. Subjects enrolled in any other interventional drug trial.
11. History of allergic reaction to compounds with similar chemical or biologic composition to imatinib.
12. Any know concurrent condition that is likely to confound investigators ability to monitor drug related adverse events.
13. Any previous treatment with any Tyrosine Kinase Inhibitor within last 90 days.
14. Any SCD related acute illness requiring hospitalization within two weeks. This will include but is not limited to:

    1. <TAB>Acute vaso-occlusive pain crisis.
    2. <TAB>Acute chest syndrome
    3. <TAB>Significant upper or lower respiratory tract infection
15. Significant upper or lower respiratory tract infection requiring hospitalization or emergency department visit within 2 weeks.
16. HIV positive subjects on Highly Active Anti-retroviral therapy (due to potential for drug interaction as well as severe immunosuppression).
17. Acute pulmonary embolism within the previous 90 days.

Subjects enrolled on this protocol who are excluded due to above criteria may proceed when their circumstances change to satisfy the exclusion criteria requirements.

Arm B (Carvedilol)

1. Current pregnancy and lactation
2. Life expectancy less than 6 months.
3. WHO functional class IV symptoms or NYHA-IV dyspnea.
4. Presence of the following medical conditions that are considered to be the cause of subject s pulmonary hypertension:

   1. <TAB>Scleroderma
   2. <TAB>Known significant obstructive or restrictive respiratory disease with FEV1, FVC or TLC below 60 percent of predicted normal.
   3. <TAB>Known diagnosis of Obesity-Hypoventilation Syndrome.
   4. <TAB>Portal hypertension or any form of severe liver dysfunction.
   5. <TAB>Structural or congenital heart disease felt to be causing the pulmonary hypertension
5. Decompensated left ventricular failure requiring intravenous inotropic therapy
6. Persistent hypotension (SBP below 90 mmHg or DBP below 50 mmHg).
7. Any subject with baseline heart rate less than or equal to 60 bpm, sick sinus syndrome, or second or third degree AV block.
8. Any initiation of new therapeutic intervention within the last 90 days or a dose change within 30 days, that is expected to have an impact on pulmonary hypertension, including but not limited to:

   1. <TAB>Specific pulmonary hypertension medication (e.g. prostacyclin analogues, endothelin receptor antagonists or phosphodiestrase-5 inhibitors)
   2. <TAB>Hydroxyurea
   3. <TAB>Scheduled blood transfusions or exchange transfusions
9. Any acute or chronic, physical or psychiatric impairment, likely to limit subject s ability to comply with study requirements as determined by investigators.
10. Subjects enrolled in any other interventional trial.
11. History of allergic reaction to compounds with similar chemical or biologic composition to carvedilol
12. Any know concurrent condition that is likely to confound investigators ability to monitor drug related adverse events
13. Use of beta-blockers within previous 90 days.
14. Cardiac index < 1.8 l/ min (2)
15. Severe renal insufficiency (creatinine clearance <30 ml/min/m(2))
16. Any SCD related acute illness requiring hospitalization within two weeks. This will include but is not limited to:

    1. <TAB>Acute vaso-occlusive pain crisis.
    2. <TAB>Acute chest syndrome
    3. <TAB>Significant upper or lower respiratory tract infection requiring hospitalization or emergency department visit
17. Significant upper or lower respiratory tract infection requiring hospitalization or emergency department visit within 2 weeks.
18. HIV positive subjects on Highly Active Anti-retroviral therapy due to potential for drug interaction.
19. Subjects with active hepatitis infection as the monitoring of drug related liver toxicity will be confounded.
20. Acute pulmonary embolism within the previous 90 days.
21. Liver function abnormalities (screening serum ALT>5 times upper limit)
22. Subjects with severe asthma as defined by presence of one or more of the following:

<TAB>- Presence of asthma symptoms throughout the day

<TAB>- Nocturnal symptoms every night

<TAB>- Need for rescue medications several times per day

<TAB>- Two or more acute exacerbations of asthma requiring systemic steroids therapy within the preceding year

<TAB>- A reduced FEV1/FVC ratio or FEV1 below 60 percent of predicted normal.

Subjects enrolled on this protocol that are excluded due to above criteria may proceed when their circumstances change to satisfy the exclusion criteria requirements.

Arm C (Hyperdynamic)

1) There are no exclusion criteria.

Arm D

1) There are no exclusion criteria.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-03-02; Primary Completion 2012-12-11 (Actual); Study Completion 2012-12-11 (Actual)

PRIMARY OUTCOMES:
An open-label non-controlled pilot study, to determine the safety and tolerability of 24-weeks of oral imatinib in SCD associated PAH and of oral carvedilol therapy in SCD associated PVH.

SECONDARY OUTCOMES:
Assess the efficacy and impact of imatinib and carvedilol on maximum exercise capacity as measured by peak oxygen consumption during a maximal CPET in SCD-PH subjects.
Assess toxicity associated with concurrent use of study drugs and hydroxyurea.
To determine appropriate monitoring, visit frequency and intensity, and to select a subject population and develop projections of statistical power for clinical efficacy endpoints.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory J Kato, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)

REFERENCES:
- [Background] Califf RM, Mark DB. Our vision for the American Heart Journal. Am Heart J. 1997 Jan;133(1):137-8. doi: 10.1016/s0002-8703(97)70261-8. No abstract available. PMID 9006304
- [Background] Sachdev V, Machado RF, Shizukuda Y, Rao YN, Sidenko S, Ernst I, St Peter M, Coles WA, Rosing DR, Blackwelder WC, Castro O, Kato GJ, Gladwin MT. Diastolic dysfunction is an independent risk factor for death in patients with sickle cell disease. J Am Coll Cardiol. 2007 Jan 30;49(4):472-9. doi: 10.1016/j.jacc.2006.09.038. Epub 2007 Jan 16. PMID 17258093
- [Background] Simonneau G, Robbins IM, Beghetti M, Channick RN, Delcroix M, Denton CP, Elliott CG, Gaine SP, Gladwin MT, Jing ZC, Krowka MJ, Langleben D, Nakanishi N, Souza R. Updated clinical classification of pulmonary hypertension. J Am Coll Cardiol. 2009 Jun 30;54(1 Suppl):S43-S54. doi: 10.1016/j.jacc.2009.04.012. PMID 19555858